CLINICAL TRIAL: NCT04110886
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending-Dose Study To Investigate the Safety, Tolerability, and Pharmacokinetics of a Kappa Receptor Agonist HSK21542 in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics of HSK21542 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK21542-101
Record Dates: First submitted 2019-08-27; First posted 2019-10-01 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Pain; Chronic Pain
Keywords: Pain; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK21542 single ascending doses (Experimental)
  Interventions: Drug: HSK21542
- Placebo single dose (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK21542 — Single dose, injection, starting dose of 0.2ug escalating up to 20ug
  Arms: HSK21542 single ascending doses
Drug: Placebo — Single dose, injection matching placebo
  Arms: Placebo single dose

SUMMARY:
This is a A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending-Dose Study To Investigate the Safety, Tolerability, and Pharmacokinetics of a kappa receptor agonist HSK21542 in Healthy Volunteers.

The study will enroll approximately 50 adults. The anticipated study duration will be up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, age 18-45 years;
* BMI between 18.0-27.0 kg/m2
* Determined by investigator to be in general good health according to medical history, comprehensive physical examination;
* Understanding of the nature, significance, potential benefits and risks of the trial, understanding of the procedures and be able to provide written informed consent voluntarily ;
* Good communication with investigators, compliance with the study requirements and willingness to stay in phase I clinical trial ward as required.

Exclusion Criteria:

* Anyone who has suffered or is currently suffering from any serious diseases, that may interfere with the results of the trial;
* Determined by investigator to be abnormal with clinical significance in Physical examination, vital signs monitoring, electrocardiogram, chest radiograph, laboratory examination;
* HBsAg positive, HCV antibody positive, Treponema pallidum antibody positive, or HIV antibody positive;
* QTcF > 450ms;
* Allergic constitution;
* Intolerance of venipuncture and/or history of haemorrhage or needle fainting;
* Drug or alcohol abuse;
* Have used any prescription, over-the-counter, Chinese herbal medicine or health products within 14 days;
* Blood donation or massive bleeding within 3 months (greater than 450 mL);
* Participants in any drug clinical trial within 3 months.
* Birth planning in the next six months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Between screening and 7-9 days after dosing
  To evaluate the safety and tolerability of HSK21542 in comparison with placebo after a single injection in healthy subjects in terms of adverse events
Number of subjects with abnormal physical examination/ abnormal vital signs/ abnormal laboratory parameters | Between screening and 7-9 days after dosing
  To evaluate the safety and tolerability of HSK21542 in comparison with placebo after a single injection in healthy subjects in terms of abnormal physical examination/ abnormal vital signs/ abnormal laboratory parameters

SECONDARY OUTCOMES:
Cmax | From the start of administration to 24 hours after administration
  Maximum (peak) plasma drug concentration
Tmax | From the start of administration to 24 hours after administration
  Time to reach maximum (peak) plasma concentration following drug administration
t1/2 | From the start of administration to 24 hours after administration
  Elimination half-life
AUC0-t | From the start of administration to 24 hours after administration
  Area under the plasma concentration-time curve from time zero to time t.
AUC0-inf | From the start of administration to 24 hours after administration
  Area under the plasma concentration-time curve from time zero to infinity
CL | From the start of administration to 24 hours after administration
  Apparent total body clearance of the drug from plasma
Vd | From the start of administration to 24 hours after administration
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wabnitz, PhD, Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No